CLINICAL TRIAL: NCT06730477
Title: Based on Plasma Exosomes Combined With Multi-omics Analysis to Reveal the Trajectory of Targeted Therapy Resistance and Novel Target Intervention Therapy in Patients With EGFR Mutation in Lung Adenocarcinoma
Brief Title: Plasma Exosomes Reveal the Efficacy of Targeted Therapy in Patients With EGFR Mutation in Lung Adenocarcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Yichang Central People's Hospital (Other); Suizhou Hospital, Hubei University of Medicine (Unknown)
Responsible Party: Principal Investigator, Yang Jin, deputy dean, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XHJY20240912
Record Dates: First submitted 2024-09-12; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Lung Adenocarcinoma; EGFR Activating Mutation
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples and tumor tissues will be retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Untreated EGFR mutated lung adenocarcinoma patients: Patients diagnosed with lung adenocarcinoma with EGFR mutations for the first time.
  Interventions: Other: observational study
- Patients with EGFR-mutated lung adenocarcinoma who are responding to targeted therapy: Patients with EGFR-mutated lung adenocarcinoma treated with targeted therapy combined with or without chemotherapy as first-line therapy, and the therapeutic effect was in the response stage.
  Interventions: Other: observational study
- Patients with EGFR-mutated lung adenocarcinoma who are resistant to targeted therapy: Patients with EGFR-mutated lung adenocarcinoma treated with targeted therapy combined with or without chemotherapy as first-line therapy, and the therapeutic effect was in drug resistance stage, or disease progression.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Efficacy of targeted therapy combined with or without chemotherapy as first-line therapy in patients with EGFR-mutated lung adenocarcinoma.

SUMMARY:
The objective of this observational study is to explore the therapeutic trajectory of targeted therapy in lung adenocarcinoma patients with epidermal growth factor receptor (EGFR) mutations. The main objective is to identify potential biomarkers that can predict the efficacy of targeted therapy through plasma exosomes and to explore strategies to reverse drug resistance to targeted therapy. Biological specimens and medical imaging data will be collected from patients already receiving targeted therapy as a first-line treatment, and followed-up will be conducted to analyze prognosis based on different patterns.

DETAILED DESCRIPTION:
The medical imaging data will be collected retrospectively and prospectively, and the blood samples and tumor tissues will be collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Pathological examination confirmed lung adenocarcinoma
* No other type of tumor was present
* Common sensitive EGFR (Ex19Del L858R or combined with other sites) mutations have been identified
* Receive targeted therapy with or without chemotherapy as first-line treatment
* ≥ 18 years and ≤80 years old

Exclusion Criteria:

* History of other malignant tumors
* Irregular treatment or poor compliance
* Incomplete clinical information or lost to follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2021 to December 2026, about 500 patients with EGFR-mutated lung adenocarcinoma who receive targeted therapy with or without chemotherapy as first-line treatment will be included in this cohort study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | A two-year period after starting treatment (Regular follow-up every three months after receiving targeted therapy combined with or without chemotherapy as first-line treatment)
  The time of disease progression is evaluated according to the Response Evaluation Criteria in Solid Tumors, version 1.1.

SECONDARY OUTCOMES:
Overall survival | A three-year period after starting treatment (Regular follow-up every six months after receiving targeted therapy combined with or without chemotherapy as first-line treatment)
  The survival time after receiving targeted therapy combined with or without chemotherapy as first-line treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Union hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No